CLINICAL TRIAL: NCT01432470
Title: A Double-blind, Placebo Controlled Multi-centre Study to Evaluate the Effects of Topical Oxytocin on Vaginal Atrophy in Postmenopausal Women
Brief Title: Study of Oxytocin to Treat Vaginal Atrophy in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PepTonic Medical AB (Industry)
Responsible Party: Dan Markusson, PeP-Tonic Medical AB
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OxyPeP-001
Record Dates: First submitted 2010-08-16; First posted 2011-09-13 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Postmenopause; Vaginal Atrophy
Keywords: vaginal atrophy
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin, Intravaginal administration (Experimental)
  Interventions: Drug: Oxytocin
- Placebo, Intravaginal administration (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Gel for intravaginal use, 600 IU once per day for 2 weeks followed by 600 IU twice a week for ten weeks
  Arms: Oxytocin, Intravaginal administration
Drug: Placebo — Gel for intravaginal use of identical appearance as active substance, once per day for two weeks followed by twice a week for ten weeks
  Arms: Placebo, Intravaginal administration

SUMMARY:
Up to 50% of all postmenopausal women, experience vaginal dryness, irritation, burning, itching or discomfort, which often make sex to become difficult or painful. These symptoms combined are known as vaginal atrophy. Vaginal atrophy is a consequence of the lining tissue of the vagina becoming thinner, drier, and less elastic due to the lack of estrogen. In addition, vaginal atrophy is associated with an increased pH, which creates an environment more susceptible to infections. The mucosal epithelium shows signs of severe atrophy and cytological examination demonstrate increased number of the basal and parabasal cells and reduced number of superficial cells.

Estrogen treatment either as hormone replacement therapy or topical application is a common treatment for vaginal atrophy. However, some women experience adverse reactions such as uterine bleeding, perineal pain and breast pain and many women are also reluctant to use estrogens due to a general negative view to this topic in the society.

Oxytocin is a peptide hormone, which is normally released into the circulation via the pituitary. The most well known effects of oxytocin are its roles in female reproduction such as facilitation of birth and breast feeding. In addition, oxytocin has in vitro been shown to exert positive effects on the proliferation of human vaginal mucosal cells from postmenopausal women.

Considering the stimulatory effects of oxytocin on vaginal mucosal cell proliferation, topical application of oxytocin to the vaginal mucosa may be an approach to treat vaginal atrophy. In one previous placebo-controlled study on 20 postmenopausal women suffering from vaginal atrophy, a gel containing oxytocin for topical intra-vaginal administration was applied daily for seven days. The results indicated that for subjects receiving topical oxytocin the vaginal atrophy assessed by histological examination was reversed after treatment. A similar effect was not seen in the placebo group, which indicated a difference between placebo and active treatment. However, the limited number of exposed subjects in this pilot study necessitates a larger study in order to generate conclusive proof of concept data for the effects of oxytocin on vaginal atrophy.

Due to the limitations of estrogens in the treatment of vaginal atrophy, many postmenopausal women are left without an effective remedy. Hence, there is a need for alternative non-estrogenic treatments of this indication. The present study is aiming to investigate the efficacy of topical oxytocin in the treatment of vaginal atrophy.

The main objective of this study is to investigate if topical oxytocin can reverse vaginal atrophy, as assessed by cytological examination of the vaginal mucosal epithelium, in postmenopausal women after 12 weeks of treatment as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* at least 40 years of age
* naturally postmenopausal women, completely without menstrual bleedings for at least four years prior to screening.
* FSH plasma levels at least 40 IU/L and 17β-estradiol levels less than 70pmol/L
* Vaginal pH more than 5.0
* BMI at most 29 kg/m2
* Vaginal atrophy verified by cytological assessment of the vaginal mucosal epithelium. Vaginal atrophy is defined as at most 5% of superficial cells.

Exclusion Criteria:

* Usage of any sex steroids including phytoestrogens, hormonal intra-uterine device or herbal medicinal products with known estrogenic effects within 3 months prior to screening.
* Usage of any lubricant for intra-vaginal administration at inclusion
* Any condition that is a contraindication to treatment with sex steroids
* Vaginal bleeding of unknown origin
* Any untreated urogenital infection within 7 days prior to inclusion
* Any prior or concurrent malignant disease or endometrial hyperplasia
* Cervical cytology at least CIN 1 assessed during screening
* Clinically significant medical history (excluding medically well-controlled hypertension and hypercholesterolemia), findings from physical examinations, vital signs, cytology, histology or laboratory analyses that may interfere with the study objectives or compromise the safety of the subject as judged by the Investigator.
* Systolic Blood Pressure at least 140 mmHg or Diastolic Blood Pressure at least 90 mmHg at screening
* Participation in any other interventional clinical trial within 3 months prior to screening
* Known or suspected drug or alcohol abuse, within 12 months prior to screening
* Concurrent and diagnosed nephrologic or hepatic disorder
* Diagnosed with HIV, Hepatitis B or C
* Known or suspected allergy to any ingredient of the study product
* Incapacity to perform study procedures, as judged by the Investigator

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The Maturation Value (MV) | 12 weeks of oxytocin treatment as compared to placebo
  The MV describes the change in percentage of superficial cells (Meisels A. The Maturation Value. Acta Cytol. 1967, Jul-Aug;11(4):249)

SECONDARY OUTCOMES:
Vaginal Atrophy | 12 weeks
  Atrophy in histological biopsies is assessed by a 4-grade scale
Quality of Life | 2 and 12 weeks
  Using a standardized QoL form
The Maturation Value | 2 weeks
  Same as primary outcome but after 2 weeks treatment
Vaginal pH | 2 and 12 weeks
Concentration of Oxytocin in serum | 0-60 min after drug admin.
  The purpose of the evaluation is only to evaluate the systemic uptake. No other PK variables than the concentration are calculated.
Clinician evaluation of vaginal mucosal appearance | 2 and 12 weeks
  Evaluation of seven different features, where every feature is assessed by a 4-grade scale.
Laboratory assessments | 2 and 12 weeks
  Clinical Chemistry, Haematology, Urine analysis, Cervical cytology,Endometrial Histology
Concentration of 17 beta-estradiol in serum | 12 weeks
Vital signs | 2 and 12 weeks
  Heart rate and blood pressure

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (2):
  - Karolinska University Hospital-Huddinge, Huddinge
  - Uppsala University Hospital, Uppsala
- Northwick Park & St Marks Hospital NHS Trust, Harrow Middlesex, United Kingdom